CLINICAL TRIAL: NCT06416839
Title: Virtual Reality Fitness Program to Promote Active Lifestyle and Psychological Wellbeing
Brief Title: VR Exercise Intervention in a Workplace Setting
Acronym: VRW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: XRWorkout, Inc (Industry)
Collaborators: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: XRW001
Record Dates: First submitted 2024-05-03; First posted 2024-05-16 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Physical Inactivity; Psychological Well-Being; Work-Related Stress
Keywords: virtual reality; exercise; lifestyle factors
MeSH Terms: conditions — Sedentary Behavior; Psychological Well-Being; Occupational Stress; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VR Exercise (Experimental): This arm will use a VR exercise game that increases in frequency, intensity and duration with each week of the intervention.
  Interventions: Behavioral: VR exercise

INTERVENTIONS:
Behavioral: VR exercise — Participation in high intensity interval training delivered on a virtual reality headset over six-week period. Participants may exercise with others in the multiplayer mode and use any feature of the application.

SUMMARY:
This research study is designed to better understand how a virtual reality (VR) exercise application may influence overall physical activity and well-being. VR games can make exercise more enjoyable and interactive, which has been shown to increase engagement in physical activity. Adult participants will do a progressive exercise program and report on overall physical activity, health, and psychological wellbeing. The intervention is expected to have a positive impact on these lifestyle factors.

DETAILED DESCRIPTION:
irtual Reality (VR) fitness applications are promising interventions to promote exercise in a home setting. Multiplayer fitness games for virtual reality platforms, addresses several common challenges associated with decreased exercise adherence such as social accountability, transportation, weather, gym memberships, and self-consciousness. This study aims to assess the impact of regular usage of a commercially available virtual reality fitness application on quality of life measures, including physical activity, health, and well-being. This study will enroll healthy participants, age 18- 50 years old, and they will be issued a Quest 2 virtual reality headset and given access to the virtual reality fitness application (VRWorkout - VRW). Participants will be asked to use VRW on a regular and progressive basis over a six-week period and to complete surveys about physical activity and wellbeing over a 9-week period. The activity completed within VRW is based on participant choice. A suggested progression schedule will be provided, but not enforced. This study of healthy working individuals, is foundational to assessing whether immersive fitness applications may be used as a lifestyle intervention to increase overall physical activity and well-being.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Individuals who have been advised by a healthcare provider that they should not participate in moderate to strenuous physical activity for any reason
* Individuals with history of seizures with photosensitivity
* Individuals with diagnosis of uncontrolled metabolic disorders
* Current lice infestation
* Current eye infection
* Body Mass Index above 30 (obese)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Physical Activity Questionnaire | Weeks 1, 3, 5, 7, and 9
  This measure assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting. A higher score indicates more physical activity.
World Health Organisation- Five Well-Being Index (WHO-5) | Weeks 1, 3, 5, 7, and 9
  The WHO-5 is a short, self-administered, and positively worded 6 point scale designed to measure the level of subjective well-being over the last two weeks. A higher score indicates better well-being.
Self-Efficacy for Exercise | Week 1 and Week 9
  This 10 point scale is a self-report on 9 items of exercise self-efficacy. A higher score indicates greater self-efficacy.
36-Item Short Form Health Survey (SF-36) | Week 1 and Week 9
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. Each of the 36 questions has a yes or no answer or a linear rating scale. These measures rely upon patient self-reporting and have been widely used. A higher score indicates better health.

SECONDARY OUTCOMES:
Health and Work Questionnaire | Weeks 1, 3, 5, 7, and 9
  The Health and Work Questionnaire was developed to assess various aspects of productivity without completely relying on direct subjective estimation. It is a multidimensional measure of productivity. It consists of 24 questions, several of which were multi-part questions, comprising six subscales. High scores indicate greater productivity or health.
Job Affect Well-being Scale | Week 1 and Week 9
  The Job-related Affective Well-being Scale (JAWS) is a scale designed to assess people's emotional reactions to their job. It asks them to indicate for each of 30 emotions (20 emotions in the short form) how often they have experienced them in the past 30 days. Higher scores indicate more positive affects related to work.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Daniels, PhD, PT, Principal Investigator — University of Mississippi Medical Center; Jennifer Reneker, PhD, PT, Study Chair — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States